CLINICAL TRIAL: NCT01795287
Title: Safety of Spinal Anesthesia in Patients With Tibial Shaft Fracture: A Single-center Randomized, Controlled Trial.
Brief Title: Safety of Spinal Anesthesia in Patients With Tibial Shaft Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: kaakinen001
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Tibial Fracture
Keywords: tibial fracture; intramedullary nailing; spinal anesthesia; patient safety
MeSH Terms: conditions — Tibial Fractures | interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal anesthesia (Active Comparator): Spinal anesthesia
  Interventions: Procedure: General anesthesia; Procedure: Spinal anesthesia
- General anesthesia (Active Comparator): General anesthesia with fentanyl, propofol and rocuronium and sevoflurane
  Interventions: Procedure: General anesthesia; Procedure: Spinal anesthesia

INTERVENTIONS:
Procedure: General anesthesia — GA will be inducted by fentanyl, propofol and rocuronium. GA will be maintained by sevofluran, fentanyl and rocuronium.
Procedure: Spinal anesthesia — hyperbaric bupivacaine 10-15 mg i.t.

SUMMARY:
There is a elevated risk of acute compartment syndrome (ACS) related to tibial shaft fractures due to oedema and reduced blood flow in traumatised tissues. This may lead to lack of oxygen and even necrosis. Symptoms of ACS are severe pain, hypoaesthesia, pain during flexion of the ankle and swollen leg in clinical examination. Paralysis and lack of distal pulses are late symptoms of ACS.

Many experts think that effective relief of pain caused by regional anaesthesia (RA) may hide the symptoms of the ACS. This may be incorrect. The evidence of dangers related to RA is based on old patient-series and single case-reports. Some of these studies report the symptoms of ACS (hypaesthesia and even pain) being caused by RA. Majority of the conclusions in these studies cannot be confirmed by an expert of RA. It is also possible that there are more hemodynamic changes related to general anaesthesia (GA) which may predispose to ACS. There are no modern, randomized and controlled studies of the safety of RA in patients with tibial shaft fracture.

DETAILED DESCRIPTION:
For some of the patients RA may be even more safe than GA. According to a large meta-analysis RA reduces the risk of several complications versus GA.

* Risk of deep vein thrombosis is reduced by 44%
* Risk of pulmonary embolism is reduced by 55 %
* Risk of major bleeding is reduced by 50%
* Risk of post operative pneumonia is reduced by 39%
* Risk of post operative respiratory is reduced by 59%

It is generally thought that RA is safer than GA for example in patients with heart or pulmonary diseases. It is also known that the use of RA reduces postoperative need of opioids, which leads to improved respiratory function and reduced post operative disorientation, delirium and nausea.

Purpose of the study: Our purpose is to gain more information of the safety of RA in patients with tibial fracture. Our hypothesis is that RA is equally safe with GA.

Implementation: Research begins with a pilot study in which RA is compared with GA. There are about 65 tibial fractures operated in our centre every year. We randomize patients to GA group (n=25) and spinal anaesthesia group (n=25). We presume that RA is equally safe with GA. However, power analysis has been made presuming that RA will increase the risk of ACS. We calculated the sample size by assuming that the compartment pressure in RA group is 10 mmHg higher than in the GA group.

GA will be inducted by fentanyl, propofol and rocuronium. GA will be maintained by sevofluran, fentanyl and rocuronium. Spinal-anaesthesia will be performed by using hyperbaric bupivacaine. The dose is 10-15 mg, depending on the needs of the patient. This will maintain RA in lower extremities for 2-4 hours, which is enough to operate a tibial shaft fracture. In both study groups the post-operative pain will be treated by intravenous and peroral oxycodone and paracetamol.

Monitoring and ethics:

* Clinical examination every hour in recovery room (oedema, temperature, cutaneous sensation, distal pulses)
* Continuous pressure-measurement of anterior compartment in the operated leg for 24 hours
* Local oxygen metabolism measured by near-infrared spectroscopy in the operated leg for 24 hours

Patients will be monitored in the recovery room for 24 hours after operation. Blood tests (creatine kinase and myoglobin) will be drawn before operation, when arriving in recovery room, 6 hours and 24 hours after operation in each patient.

ELIGIBILITY:
Inclusion Criteria:

Patients with a unilateral tibial shaft fracture which needs to be operated are included.

Exclusion Criteria:

* refusal of the patient
* severe, generalized atherosclerosis
* massive obesity
* marked mental retardation, dementia
* bilateral tibial shaft fracture
* polytrauma, such as head injury
* bleeding diathesis
* aortic stenosis
* infection at the injection site
* certain medications affecting bleeding
* sepsis
* hypovolemia
* conversion to general anaesthesia due to technical difficulties
* anesthesiologist has a strong opinion towards GA/RA
* foreign patient and marked translation difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-03; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Compartment pressure | 0-24 hours after surgery
  Continuous measurement of anterior compartment pressure in the operated leg

SECONDARY OUTCOMES:
INVOS values after surgery | 0-24 hours after surgery
  Continuous monitoring of INVOS values in the anterior and postolateral position in the operated leg

CONTACTS AND LOCATIONS:
Overall Officials: Timo Kaakinen, MD, PhD, Study Director — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Lehto PM, Vakkala MA, Lantto IP, Ohtonen P, Liisanantti JH, Kaakinen TI. Spinal Anaesthesia Versus General Anaesthesia for Patients With Tibia Shaft Fractures-A Randomized Controlled Study. Acta Anaesthesiol Scand. 2025 Sep;69(8):e70111. doi: 10.1111/aas.70111. PMID 40792424